CLINICAL TRIAL: NCT05583721
Title: An Evaluation of the Relationship Between Abnormal Myocardial Perfusion and Diastolic Dysfunction in Sickle Cell Disease Using PET (Stress-Rest) Myocardial Perfusion Imaging (MYPERS)
Brief Title: Relationship Between Abnormal Myocardial Perfusion and Diastolic Dysfunction in Sickle Cell Disease Using PET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MYPERS
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease patients; Healthy controls; Abnormal diastolic heart function; Coronary Flow Reserve (CFR); Coronary microvasculature dysfunction; Myocardial perfusion reserve; Positron emission tomography (PET) imaging; PET (stress-rest) myocardial perfusion imaging
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ammonia; 1,3-(N'-amidinosulfanilamide)-2,2,2,4,4,4-hexachlorocyclodiphosph(V)azane; regadenoson; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stratum A (Experimental): Sickle Cell patients with diastolic dysfunction
  Interventions: Drug: [13N]NH3; Drug: Lexiscan; Diagnostic Test: Positron emission tomography
- Stratum B (Experimental): Sickle cell patients without diastolic dysfunction
  Interventions: Drug: [13N]NH3; Drug: Lexiscan; Diagnostic Test: Positron emission tomography
- Stratum C (Experimental): Healthy controls
  Interventions: Drug: [13N]NH3; Drug: Lexiscan; Diagnostic Test: Positron emission tomography

INTERVENTIONS:
Drug: [13N]NH3 — Ammonia N 13 (a radioactive tracer) will be given per intravenous (IV) injection for diagnostic purposes in conjunction with positron emission tomography (PET) imaging.
  Other Names: [N-13] Ammonia; azane; CAS# 34819-78-8
Drug: Lexiscan — Given IV prior to PET stress test
  Other Names: Regadenoson
Diagnostic Test: Positron emission tomography — Participants will complete a onetime PET (stress-rest) myocardial perfusion scan.
  Other Names: PET

SUMMARY:
There is limited information on what causes injury to the heart in individuals with Sickle Cell Disease (SCD). Researchers in this study want to see if decreased blood flow to the heart during stress could be causing the heart damage seen in SCD patients. They also want to test people who don't have SCD to see if their hearts react the same way under stress.

Primary Objective

* To estimate the coronary flow reserve (CFR) (also referred to as myocardial perfusion reserve), as measured by PET stress-rest myocardial perfusion imaging, in SCD patients with and without diastolic dysfunction, and healthy controls.

Secondary Objectives

* To investigate the relationship between decreased CFR (quantified with PET stress- rest myocardial perfusion imaging) and presence of abnormal diastolic parameters

DETAILED DESCRIPTION:
This study requires two visits. The first visit includes blood tests, an electrocardiogram (EKG), and an echocardiogram. The second visit includes a positron emission tomography (PET) stress test and a blood test.

Subjects will be considered off-study one week after all post PET imaging study tests have been completed along with the next day and one-week follow-up phone calls are completed.

ELIGIBILITY:
Inclusion Criteria - Stratum A: Sickle cell patients with diastolic dysfunction

* 18 to 21 years of age
* Black
* Diagnosis of SCD of HbSS and HbSβ0thalassemia genotypes
* Three or more abnormal diastolic parameters (based on guidelines by American Society of echocardiography)

Inclusion Criteria - Stratum B: Sickle cell patients without diastolic dysfunction

* 18 to 21 years of age
* Black
* Diagnosis of SCD of HbSS and HbSβ0thalassemia genotypes
* Two or less abnormal diastolic parameters

Inclusion Criteria - Stratum C: Healthy controls

* 18 to 21 years of age
* Black
* Two or less abnormal diastolic parameters

Exclusion Criteria - Stratum A:

* Recent hospitalization for vaso-occlusive pain crisis or acute chest syndrome in last 4 weeks
* Blood transfusion in the last 3 months
* Individuals with signs, symptoms or EKG findings of acute myocardial ischemia, infarction or unstable angina
* Individuals with history of VT/VF or SVT
* Previous cardiac surgery
* Known congenital heart disease (other than patent ductus arteriosus or Atrial septal defect)
* Stenotic valvular disease or left main coronary artery stenosis
* History of myo/pericarditis
* Left ventricle systolic dysfunction
* Cardiovascular instability/uncontrolled hypertension (h/o hypertensive urgency or emergency)
* History of sinus node dysfunction or high grade AV nodal block
* History of aborted sudden cardiac death or cardiac arrest
* Current seizure disorder on AED
* Pregnant/Breast-feeding
* Any medical or social reason, which, in the opinion of the principal investigators would make the participation of the subject ill-advised.

Exclusion Criteria - Stratum B:

* Diagnosed with three or more abnormal diastolic parameters (based on guidelines by American Society of echocardiography)
* Recent hospitalization for vaso-occlusive pain crisis or acute chest syndrome in last 4 weeks
* Blood transfusion in the last 3 months
* Individuals with signs, symptoms or EKG findings of acute myocardial ischemia, infarction or unstable angina
* Individuals with history of VT/VF or SVT
* Previous cardiac surgery
* Known congenital heart disease (other than patent ductus arteriosus or Atrial septal defect)
* Stenotic valvular disease or left main coronary artery stenosis
* History of myo/pericarditis
* Left ventricle systolic dysfunction
* Cardiovascular instability/uncontrolled hypertension (h/o hypertensive urgency or emergency)
* History of sinus node dysfunction or high-grade AV nodal block
* History of aborted sudden cardiac death or cardiac arrest
* Current seizure disorder on AED
* Pregnant/Breast-feeding
* Any medical or social reason, which, in the opinion of the principal investigators would make the participation of the subject ill-advised.

Exclusion Criteria - Stratum C:

* All genotypes of SCD
* Diagnosed with three or more abnormal diastolic parameters (based on guidelines by American Society of echocardiography)
* Anemia of grade 2 or worse (per CTCAE v5.0) at study visit 1
* Individuals with signs, symptoms or EKG findings of acute myocardial ischemia, infarction or unstable angina
* Individuals with history of VT/VF or SVT
* Previous cardiac surgery
* Known congenital heart disease (other than patent ductus arteriosus or Atrial septal defect)
* Stenotic valvular disease or left main coronary artery stenosis
* History of myo/pericarditis
* Left ventricle systolic dysfunction
* Cardiovascular instability/uncontrolled hypertension (h/o hypertensive urgency or emergency)
* History of sinus node dysfunction or high-grade AV nodal block
* History of aborted sudden cardiac death or cardiac arrest
* Current seizure disorder on AED
* Pregnant/Breast- feeding
* Any medical or social reason, which, in the opinion of the principal investigators would make the participation of the subject ill-advised.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Mean and standard deviation of coronary flow reserve (CFR) | Visit 2, approximately 4 weeks after study entry (procedure takes approximately one hour)
  We will estimate the mean and standard deviation of CFR, as measured by PET myocardial blood flow reserve imaging, in young adult SCD patients with and without diastolic dysfunction and healthy controls.
CFR difference among Stratum A, Stratum B, and Stratum C | Visit 2, approximately 4 weeks after study entry (procedure takes approximately one hour)
  We will compare whether the CFR is different among 3 predefined strata: Stratum A; SCD with diastolic dysfunction patients , Stratum B; SCD without dysfunction patient control, and Stratum C; normal healthy controls by one-way ANOVA or Kruskal-Wallis one-way analysis of variance, depending on the distribution of the data. If the difference exists, the pairwise comparison will be carried out by two sample t test or Wilcoxon rank sum test between two strata.

SECONDARY OUTCOMES:
Relationship between decreased CFR (quantified with PET stress-rest myocardial perfusion imaging) and presence of abnormal diastolic parameters | Visit 2, approximately 4 weeks after study entry (procedure takes approximately one hour)
  The following is the grouping of diastolic parameters used in this study: Group 1: 0 or any 1 diastolic variable abnormal; Group 2: Any 2 variables abnormal; Group 3: Any 3 or more variables abnormal . We will first summarize the mean and standard deviation CFR values for each diastolic group. One-way ANOVA or Kruskal-Wallis one-way ANOVA will be used to explore whether there are any statistically significant differences between the means of these three groups. If a difference exists, the pairwise comparison will be carried out by two sample t test or Wilcoxon rank sum test between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Parul Rai, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols